CLINICAL TRIAL: NCT05488184
Title: Pilot Study to Evaluate the Organoleptic Perception of an Specific Oral Nutritional Supplements for Oncological Patients
Brief Title: Study to Evaluate the Organoleptic Perception of Oral Nutritional Supplements for Oncological Patients
Acronym: SENSORIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Adventia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HULP 5254
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2019-09

CONDITIONS: Cancer; Nutrition Related Cancer; Malnutrition
Keywords: cancer; nutrition; oral nutrition supplement; organoleptic properties; pilot study
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Supplement (Experimental): Five different flavours of Oral Nutritional Supplement (ONS) prototypes were tested: tropical, pineapple, brownie, ham, tomato
  Interventions: Dietary Supplement: Flavoured Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Dietary Supplement: Flavoured Oral Nutritional Supplement (ONS) — Sensory analysis of different ONS of sweet (pineapple, tropical, brownie) and acid flavoured (tomato, ham)
  Other Names: Experimental

SUMMARY:
Nutritional therapy is key to helping cancer patients get the nutrients they need to maintain body weight, strength, tissue and organ integrity, and face likely infections. Some cancer treatments work best when the patient is well nourished and has enough calories and macronutrients from food. According to the latest consensus, the first step in nutritional intervention is nutritional recommendations or dietary advice. These recommendations must be realized if the patient is capable of ingesting at least 75% of the nutritional requirements that correspond to them and, if there is no approach to an upcoming risk therapy. As long as the oral route is not damaged, in dietary advice this should always be the first option. Increasingly, laboratories specialized in nutritional products prepare and improve the composition of supplements. They are complete, specific and perfect to meet the dietary needs of patients who require it. But, to fulfill their function, they have to be ingested by people and for that they have to have good organoleptic characteristics, a very important nuance that is sometimes not taken into account in the manufacture of these products. It is the object of Adventia Pharma, S.L. develop new Oral Nutritional Supplements specific for cancer patients and that meet optimal organoleptic characteristics. For this reason, a pilot study will be carried out that will evaluate different sensory and organoleptic aspects of the prototypes of supplements developed by the company to determine the consumer's reaction to the products developed and subsequently be able to select the one with the greatest acceptance.

DETAILED DESCRIPTION:
In cancer patients there is great difficulty in maintaining and/or improving their nutritional status if early nutritional support or surveillance measures are not taken, which can prevent progressive deterioration. The act of eating in a traditional way influences the perception of normality or illness in patients. Nutrition not only represents an essential parameter in the development of cancer, but it can also be a fundamental factor in its treatment. In the case of cancer, both the disease and the treatment have a direct impact on nutrition and generate bodily changes that gradually appear as a consequence of them. Cancer produces a direct decrease in intake, due to the disease, the metabolic alteration induced by the tumor, the physiological changes produced, the effects of cancer treatment and the presence of symptoms (depression, anorexia, vomiting, diarrhoea, pain , etc.); mechanically interfering with the normal transit of the digestive tube, or indirectly through the secretion of substances that act on peripheral receptors or on the hypothalamus. The patient may therefore be faced with a tumor cachexia syndrome characterized by weight loss, reduced fat and muscle mass, anorexia with reduced intake, early satiety, hypoalbuminemia, anemia, and progressive weakness, among others. others. This malnutrition aggravates the problem of immunosuppression that the patient already has due to his cancer, and has a great impact on functional capacity, with an increase in complications, the rate of infections, decreases tolerance to cancer treatment, the patient's quality of life and thus their chances of survival.

Oral nutritional support consists of the administration of nutrients and other necessary adjuvant therapeutic substances, with the purpose of improving or maintaining the nutritional status of a patient. This support is indicated for patients who are in different clinical situations such as limitation of intake, swallowing, transit, digestion, absorption and/or metabolism of nutrients, or who have special energy and/or nutrient requirements that cannot be covered with natural food.

Therefore, the main objectives of nutritional supplementation in cancer patients are the following:

* Prevent or correct nutritional deficiencies.
* Minimize the side effects of anti-neoplastic treatment.
* Improve tolerance to anti-neoplastic treatment.
* Improve Life Quality.
* Help achieve optimal body weight.
* Educate the patient/family about special nutritional needs. In conclusion, the choice of a nutritional supplement if it is indicated for a specific nutritional treatment should be based on its composition, its physical characteristics (taste, smell, texture...) and the underlying disease. It should also be adjusted as far as possible to the patient's tastes. There are different types of formulas, some designed with specific nutrients for certain diseases, disorders or conditions (oncology, pressure ulcers, constipation, diarrhea, etc.) and others that are intended for patients without specific needs.

Increasingly, laboratories specialized in nutritional products prepare and improve the composition of supplements. They are complete, specific and perfect to meet the dietary needs of patients who require it. But, to fulfill their function, they have to be ingested by people and for that they have to have good organoleptic characteristics, a very important nuance that is sometimes not taken into account in the manufacture of these products.

For this reason, a randomized, cross-sectional and double-blind pilot study was performed to evaluate different organoleptic properties of 5 oral nutritional prototype of supplements. The investigators included 30 patients. Each volunteer tasted the 5 different prototypes the same day in a different order.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 years old.
* Patients diagnosed with cancer (any type) and who have started or are going to start with chemo and/or radiotherapy treatment with or without surgery.
* Adequate cultural level and understanding
* Agree to participate in the study

Exclusion Criteria:

* Subjects with severe infection or major surgery in the previous three months.
* Subjects with an infectious process at the time of the study.
* Subjects with insulin dependent diabetes.
* Subjects with dementia, mental illness or decreased cognitive function.
* Pregnant or breastfeeding women.
* Subjects with body mass index ≥ 40kg/m2.
* Subjects who rejects oral nutritional supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Color of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.
Taste of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.
Flavor of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.
Aftertaste of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.
Texture of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.
Thickness of the experimental ONS | Day 1
  It will be evaluated through an Organoleptic Hedonic Scale that will measure 5 levels, to which a score will be associated: I dislike it a lot (1 point); I dislike it moderately (2 points); I neither like nor dislike (3 points); I like it moderately (4 points); I like it a lot (5 points). The minimum score of the questionnaire is 6 points, while the maximum is 30.

SECONDARY OUTCOMES:
Weight (kg) | Day 1
  It is measured using a digital scale for clinical use (capacity 0-150 kg), with the person positioned with their back to the viewer, without shoes, wearing a minimum of warm clothing (pants and t-shirt), heels together, looking forward and posture straight body.
Waist circumference (cm) | Day 1
  The subject assumes a position with arms crossed at the chest. The perimeter is taken at the narrowest level, between the lower costal margin (10th rib) and the iliac crest. The anthropometrist stands in front of the subject, who has his arms slightly abducted, to allow the waist to run around the abdomen. Values greater than 80 centimeters (women) and 94 centimeters (men) are considered a risk for cardiovascular diseases.
Body Mass Index (kg/m2) | Day 1
  It is the relationship between the individual's body weight (kg) and height (m) squared: Weight/Height2. Values greater than 24,9 kg/m2 are considered as overweight
24 hour food record questionnaire | Day 1
  Questionnaire to find out the nutritional and dietary habits of each participant. The volunteer will write down all the food and drinks ingested in the previous day of clinical visit (24 hours). The answers will allow calculating the total amount of food consumed and calories ingested. In addition, the data will be evaluated quantitatively and qualitatively, classifying the diet in terms of diversity and balance following the recommendations of the Spanish Society of Community Nutrition (SENC 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Marina Morato Martínez, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Bricia Lopez Plaza, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No